CLINICAL TRIAL: NCT02347670
Title: Comparison Study of Glaucoma Eye Care Follow-Up Adherence in a High Risk Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Partridge Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB#14-380
Record Dates: First submitted 2014-12-05; First posted 2015-01-27 (Estimated); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1M- Community Site (Active Comparator): Participants randomized to Group 1-Main will attend follow-up visits at one of the four main community sites. A glaucoma specialist will perform the comprehensive eye examination and a ophthalmic technician will conduct the testing. There will be no charge or co-pay for these visits. Group 1 participants will test the efficacy of the patient navigator to improve follow-up adherence. During the first and final follow-up visit, those enrolled will undergo the National Eye Institute-Visual Function Questionnaire-25 and the Geriatric Depression Scale-15 and Research Participation Questionnaire.
  Intervention: Efficacy-patient navigator to improve follow-up adherence
  Interventions: Behavioral: Efficacy-patient navigator to improve follow-up adherence
- Group 2- Office-Based (Active Comparator): Office-Based, Follow-Up Eye Care with Patient Navigation Protocol: Participants randomized to Group 2 will attend follow-up visits at the Wills Eye Hospital Glaucoma Research Center. A glaucoma specialist will perform the eye examination. Ophthalmic technicians will conduct the testing. There will be no charge or co-pay for these visits. Group 1 participants will test the efficacy of the patient navigator to improve follow-up adherence. During the first and final follow-up visit, those enrolled will undergo the National Eye Institute-Visual Function Questionnaire-25 and the Geriatric Depression Scale-15 and Research Participation Questionnaire.
  Intervention: Efficacy-patient navigator to improve follow-up adherence
  Interventions: Behavioral: Efficacy-patient navigator to improve follow-up adherence
- Group 3- Office-Based (Active Comparator): Group 3- follow-up eye care at the Wills Eye Hospital. There will be no charge or co-pay for these visits. Those enrolled will undergo the National Eye Institute-Visual Function Questionnaire-25 and the Geriatric Depression Scale-15 and Research Participation Questionnaire. These participants will receive a phone number to call and schedule their appointment and will receive a reminder phone call similar to the standard appointment-reminding procedure commonly used at the Wills Eye Hospital. Group 3 represents a realistic choice currently available for patients and thus will be used to compare with usual care and will have 2-3 visits over the one-year period depending on diagnosis.
  Intervention: Office-Based Usual Care
  Interventions: Behavioral: Office-Based Usual Care
- Group 1R- Community Site (Active Comparator): Participants randomized to Group 1-Randomized will attend follow-up visits at one of the four main community sites, these participants were randomized from the 40 community sites to the closest community location. A glaucoma specialist will perform the comprehensive eye examination. Ophthalmic technicians will conduct the testing. There will be no charge or co-pay for these visits. Group 1 participants will test the efficacy of the patient navigator to improve follow-up adherence. During the first and final follow-up visit, those enrolled will undergo the National Eye Institute-Visual Function Questionnaire-25 and the Geriatric Depression Scale-15 and Research Participation Questionnaire.
  Intervention: Efficacy-patient navigator to improve follow-up adherence
  Interventions: Behavioral: Efficacy-patient navigator to improve follow-up adherence

INTERVENTIONS:
Behavioral: Efficacy-patient navigator to improve follow-up adherence — Over the course of 1 year, a 6-person team comprised of one attending physician ; ophthalmic technicians, project managers/community health educators , and patient navigators will complete a baseline eye examination visit, baseline assessment, and 2-3 follow-up visits. The equipment will occupy a designated location at each site for 1 to 2 days, from 9 a.m. to 3 p.m., with at least 15 eye examinations performed each day. With assistance from the patient navigator, participants will receive assistance with scheduling appointments, arranging transportation, reminder letters, and referral s for ocular care.
  Arms: Group 1M- Community Site; Group 1R- Community Site; Group 2- Office-Based
Behavioral: Office-Based Usual Care — Over the course of 1 year, a 6-person team comprised of one attending physician ; ophthalmic technicians, project managers/community health educators , and patient navigators will complete a baseline eye examination visit, baseline assessment, and 2-3 follow-up visits. The equipment will occupy a designated location at each site for 1 to 2 days, from 9 a.m. to 3 p.m., with at least 15 eye examinations performed each day.
  This intervention group will receive a phone number to schedule an appointment. Participants in the usual-care group who have scheduled an appointment will receive an automated phone call similar to the standard appointment-reminding procedure used at the Wills Eye Hospital.
  Arms: Group 3- Office-Based

SUMMARY:
The project aims to determine the effectiveness of a patient-centered health care delivery system focused on improving follow-up adherence in patients diagnosed with glaucoma. Over the course of 1 year, a 6-person team comprised of one attending physician; project managers and community health educators, ophthalmic technician, and patient navigators will complete a baseline visit, baseline assessment and 2-3 follow-up visits. The patient navigator will assist participants in community groups and a portion of the office-based participants with scheduling follow-up appointments

DETAILED DESCRIPTION:
The Partridge Foundation has funded the Wills Eye Hospital Glaucoma Research Center for the project: Comparison Study of Glaucoma Eye Care Follow-up Adherence in a High-Risk Population to continue follow-up eye care for those who received a glaucoma diagnosis during the 2010 Center for Disease Control and Prevention funded cooperative agreement: Improving Access to Eye Care among High-Risk Persons for Glaucoma in Philadelphia Project. The project aims to determine the effectiveness of a patient -centered health care delivery system focused on improving follow-up adherence in patients diagnosed with glaucoma.

There are approximately 700 potentially eligible persons from the 39 community sites, and of that the investigators hope to enroll 250 into 1 of four groups. Eligible participants have participated in the community-based comprehensive eye examination, have received a diagnosis of glaucoma-suspect or any type of glaucoma, including open angle glaucoma, chronic angle closure glaucoma, ocular hypertension, anatomically narrow-angle, pigmentary glaucoma, low tension glaucoma, or pseudoexfoliative glaucoma (identified using International Classification of Diseases (ICD)-9 codes), are recommended for follow-up care and have attended their Center for Disease Control and Prevention 6-month follow-up visit, are willing and able to give informed consent and participate for 1 year, any have undergone laser therapy. Excluded subjects are unwilling to attend randomized site for follow-up visits or prefers to continue follow-up eye care with their personal ophthalmologists.

Over the course of 1 year, a 6-person team comprised of one attending physician; project managers and community health educations, ophthalmic technician, and patient navigators will complete a baseline visit, baseline assessment and 2-3 follow-up visits in community and office-based locations. A leased Wills Eye van will transport the intervention team and all necessary equipment to the site. The equipment will occupy a designated location at each site for 1 to 2 days per month, from 9 a.m. to 3 p.m., with at least 15 eye examinations performed each day. The same team will see participants who are randomized to the Wills Eye Glaucoma Research Center location.

Participants randomized to receiving help in patient navigation protocol at the community and office-based locations will receive more individualized care than others such as assistance with scheduling; a confirmation letter, text or email; a personal phone call the day before the appointment; and assistance with rescheduling appointments as needed and will consistently arrange transportation to appointments as needed, provide materials, and accompany study participants to their follow-up appointments at Wills Eye. Patient navigators, ocular technicians, and physicians will also communicate with family members regarding recommended follow-up visits, medication refills, and laser-therapy recommendations, as needed.

Participants randomized to usual care protocol at the office-based location will receive a phone number to call and schedule an appointment. Prior to the follow-up visit, participants in the usual-care group who have scheduled an appointment will receive an automated phone call similar to the standard appointment-reminding procedure commonly used at the Wills Eye Hospital. If participants do not show-up for their appointment that will be documented. Participants in the usual-care group will receive any necessary interpretation services, educational materials, and referrals to cataract surgery or other eye-care services, as needed. The intervention team will assure that participants with literacy issues can understand all information. This group is a realistic choice currently available for patients and thus will be used to compare with the patient navigator protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the Wills Eye community-based comprehensive eye examination.
* Have a diagnosis of glaucoma-suspect or any type of glaucoma, including open angle glaucoma, chronic angle closure glaucoma, ocular hypertension, anatomically narrow-angle, pigmentary glaucoma, low tension glaucoma, or pseudoexfoliative glaucoma (identified using ICD-9 codes).
* Are recommended for follow-up care.
* Are willing and able to give informed consent and participate for 1 year.
* May have undergone laser therapy.

Exclusion Criteria:

* Are unwilling to go to any site for follow-up visits.
* Requested to follow-up only with their own ophthalmologist for their glaucoma eye-care.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of Patient Navigator in a community setting or office based setting or usual care | Following 1 year
  Using data from randomized patients only, we will fit population average Poisson regression models using generalized estimating equations to estimate the rates of timely attendance by randomization assignment and assess the efficacy of the interventions while accounting for within-site clustering. The primary analysis will be adjusted for baseline individual characteristics believed to be associated with adherence to follow-up including age, glaucoma diagnosis, geriatric depression score, and overall vision-related quality of life.

SECONDARY OUTCOMES:
Differences between rates of follow-up adherence; Community Groups (1-Main v.s Group 1-Randomized). | 1 Year
  This analysis will be primarily descriptive since although we expect follow-up to be higher in Group 1-Main (Main Community Group), we do not expect the difference to be large.
Effectiveness of the patient navigator intervention on long-term patterns of follow-up. | 1 Year
  Additional secondary analysis will consider the effect of intervention on long-term patterns of follow-up. Since the pattern of expected visits differs by severity, we will classify subjects as long-term adherent if they attend all of their recommended follow-up visits and non-adherent otherwise. Analysis will use the same model as the primary outcome analysis.

OTHER OUTCOMES:
Differences of baseline patient characteristics of glaucoma severity, vision-related quality of life, and depression. | 1 year
  We will consider whether the effect of the intervention differs by baseline patient characteristics of glaucoma severity, vision-related quality of life, and depression. The primary model will be extended to include the interaction between these variables and randomization assignment to allow for estimation of intervention effects by baseline categories.

CONTACTS AND LOCATIONS:
Overall Officials: L. J. Katz, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A manuscript has been published.

REFERENCES:
- [Background] Hark LA, Johnson DM, Berardi G, Patel NS, Zeng L, Dai Y, Mayro EL, Waisbourd M, Katz LJ. A randomized, controlled trial to test the effectiveness of a glaucoma patient navigator to improve appointment adherence. Patient Prefer Adherence. 2016 Sep 8;10:1739-48. doi: 10.2147/PPA.S108391. eCollection 2016. PMID 27660423